CLINICAL TRIAL: NCT05595421
Title: Clinical and Electrophysiological Outcomes of Transcranial Direct Current Stimulation in Patients With Treatment Resistant Obsessive Compulsive Disorder
Brief Title: Clinical and Electrophysiological Outcomes of tDCS in Patients With Treatment Resistant OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-An Chang, MD, Professor, Attending Psychiatrist, Department of Psychiatry, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-108-03-001
Record Dates: First submitted 2022-10-22; First posted 2022-10-27 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; treatment resistance; EEG; transcranial direct current stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: A three arm/group parallel interventional study model.
Who Masked: Outcomes Assessor
Masking Description: Study outcomes are measured by clinical raters blinded to the arms and interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The right cerebellum (anode) and the left OFC (cathode) tDCS (Experimental): Stimulation sessions will be carried out using a neuroConn DC stimulator (Ilmeneau, GmbH) with two rubber electrodes placed inside two 5 × 7 cm (35 cm2) sponge electrodes soaked in a saline solution (0.9% NaCl). Electrodes will be placed on the basis of the international 10-20 electrodes placement system. The cathode will be placed over the left OFC on the FP1 point according to the EEG international reference. The anode will be placed over the right cerebellum 3 cm below the inion and 1 cm right from the midline. Patients will receive twice-daily sessions separated by at least 1 h for 10 consecutive weekdays. One session of tDCS consists in delivering a direct current of 2 mA during 20 min.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- The bilateral pre-SMA (cathode) and right deltoid (reference) tDCS (Experimental): Stimulation sessions will be carried out using a neuroConn DC stimulator (Ilmeneau, GmbH). The stimulator is connected to two rubber electrodes which are placed inside two sponge electrodes soaked in a saline solution (0.9% NaCl), respectively. The active electrode (cathode) is 5×5 cm and placed on the sagittal midline at 15% of the distance between inion and nasion anterior to Cz (vertex), using the International 10-20 EEG System, to target the bilateral presupplementary motor area (pre-SMA). The reference electrode is 5×7 cm and placed on the lateral surface of the patient's right deltoid. Patients will receive twice-daily sessions separated by at least 1 h for 10 consecutive weekdays. One session of tDCS consists in delivering a direct current of 2 mA during 20 min.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- The left OFC (cathode 1), bilateral pre-SMA (cathode 2), and right deltoid (reference) tDCS (Experimental): Stimulation sessions are carried out using a neuroConn DC stimulator (Ilmeneau, GmbH). The stimulator is connected to a 2 × 1 wire adaptor (Equalizer Box, NeuroConn) that links three rubber electrodes placed inside sponge electrodes soaked in a saline solution (0.9% NaCl) will be applied. One active electrode (the 1st cathode) is 5×5 cm and placed on the sagittal midline at 15% of the distance between inion and nasion anterior to Cz (vertex), using the International 10-20 EEG System, to target the bilateral presupplementary motor area (pre-SMA). The other active electrode (the 2nd cathode) is 5×7 cm and placed over the left OFC on the FP1 point according to the EEG international system. The reference electrode is 5×7 cm and placed on the lateral surface of the patient's right deltoid. Patients will receive twice-daily sessions separated by at least 1 h for 10 consecutive weekdays. One session of tDCS consists in delivering a direct current of 2 mA during 20 min.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — See detail in arm/group descriptions regarding the intervention.

SUMMARY:
The aim of this study is to analyze the effectiveness of three different montages of transcranial direct current stimulation (tDCS) in treating treatment-resistant OCD.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) typically starts between childhood and early adulthood and is characterized by the presence of obsessions and/or compulsions and a typically chronic clinical course. Around one-third of OCD patients fail to benefit significantly from first-line treatment, e.g., serotonin reuptake inhibitors (SRIs) or cognitive behavioral therapy (CBT). Combining, augmenting, and switching strategies as second-line treatments also fail to bring much benefit to these patients. When the first-line and second-line treatments fail, alternative treatments (e.g., non-invasive brain stimulation techniques) should be considered. A proposed pathophysiology of OCD is the dysfunction of cortico-striato-thalamo-cortical circuitry including the medial prefrontal cortex [i.e., supplementary motor area (SMA) and anterior cingulate cortex (ACC)], the dorso-lateral prefrontal cortex (DLPFC), the orbitofrontal cortex (OFC), and the basal ganglia. Among novel therapeutic options of non-invasive brain stimulation, transcranial direct current stimulation (tDCS) has shown positive results (e.g., cathodal tDCS over the pre-SMA, tDCS with the cathode over the left OFC and the anode over the right cerebellum, and tDCS with anode over Pre-SMA and cathode over right supra-orbital area) in treatment-resistant OCD. However, there is unclear evidence regarding the best tDCS montage for treatment-resistant OCD. This study investigates the effects of three different tDCS montages in reducing the symptoms of patients with treatment-resistant OCD. Eligible participants with treatment-resistant OCD will be allocated randomly into three groups of different tDCS montages [1. The right cerebellum (anode) and the left OFC (cathode) tDCS; 2. The bilateral pre-SMA (cathode) and right deltoid (reference) tDCS; 3. The left OFC (cathode 1), bilateral pre-SMA (cathode 2), and right deltoid (reference) tDCS]. Patients will receive twice-daily sessions separated by at least 1 h for 10 consecutive weekdays. One session of tDCS consists in delivering a direct current of 2 mA during 20 min. The primary outcome is the difference in the change of the score of the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) between three different montages of tDCS. Electrical activity of the brain as measured by EEG, autonomic function as measured by heart rate variability, and cognitive functioning as secondary outcomes will be measured before and after three different montages of tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants aged 20-65 with the primary clinical diagnosis of DSM-5-defined obsessive-compulsive disorder.
* Being treatment-resistant, as revealed by a Yale-Brown Obsessive and Compulsive Scale score (Y-BOCS) >16 despite at least two selective serotonin reuptake inhibitor (SSRI) trials of adequate dose and duration (or refusal to take medication for personal choice) and having been offered prior cognitive behavior therapy (CBT) by a trained practitioner.
* The dosages of undergoing psychopharmacological medications having remained unchanged for 1 month before the beginning of the trial and remaining unchanged throughout the entire duration of the study.
* Agreement to participate in the study and provide the written informed consent.

Exclusion Criteria:

* Having contraindications for transcranial electrical stimulation or transcranial magnetic stimulation, e.g., pacemakers, metallic or magnetic pieces in the head/brain, ear implants and other implantable brain medical devices.
* Pregnancy or breastfeeding at enrollment.
* Having active substance use disorder (in exception to caffeine and/or tobacco).
* Having a history of seizures.
* Having a history of intracranial neoplasms or surgery, or a history of severe head injuries or cerebrovascular diseases.
* Skin lesions on scalp at the area of electrode application.
* Having unstable medical conditions at enrollment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The change over time in the score of the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups) | Six weeks
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a 10-item scale designed to measure the severity and type of symptoms in people with obsessive-compulsive disorder (OCD) over the past seven days. The symptoms assessed are obsessions and compulsions. Total Y-BOCS scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms. Scores on the obsession and compulsion subscales range from 0 to 20, but only the total Y-BOCS score is interpreted.

SECONDARY OUTCOMES:
The change over time in the score of self-reporting OCD Visual Analog Scale (OCD-VAS) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups) | Six weeks
  The participants use the self-reporting OCD Visual Analog Scale (OCD-VAS) to rate on a 10-point scale the current obsessive and compulsive symptoms (0 = Feel Worst Ever to 10 = Feel Best Ever).
The change over time in the score of the Clinical Global Impression improvement (CGI-I) subscales of the CGI-S (severity scale) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups) | Six weeks
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Clinicians ask: "Compared to the patient's condition at baseline, this patient's average condition is rated as from 1 (Very much improved) to 7 (Very much worse).
The change over time in the score of Hamilton Depression Rating Scale (HAM-D) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups) | Six weeks
  The HAMD is designed to be administered by a trained clinician, and it contains 17 items rated on either a 3- or 5-point scale, with the sum of all items making up the total score. Low scores indicate less depression severity and greater function.
The change over time in the score of Hamilton Anxiety Rating Scale (HAM-A) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups) | Six weeks
  The total score of HAMA ranges from 0-56, with each of the 14 items being scored on a severity scale of 0 to 4. Low scores indicate less anxiety severity and greater function.
The change over time in the score of the Taiwanese version of World Health Organization Quality of Life-BREF (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups) | Six weeks
  The Taiwanese version of World Health Organization Quality of Life-BREF is a self-report 28 items (2 generic, 7 Physical, 6 Psychological, 4 Social, and 9 Environment items) questionnaire. Item scores range from 1 (the worst condition) to 5 (the best condition), except for 3 items (Ph1, Ph2, and Ps6), which are reverse coded. A higher score indicates better quality of Life.
The changes over time in the results of Continuous Performance (CPT, version 2.0) (from baseline to the end of intervention) | Two weeks
  A neuropsychological test that examines the performance of prefrontal-mediated task
The changes over time in the results of Color Trails Test (CTT) (from baseline to the end of intervention) | Two weeks
  The CTT, a culture-neutral version of the Trail Making Test, was selected to measure sustained visual attention. The CTT consists of two parts (CTT-1 and CTT-2). The CTT-1 requires participants to connect a series of numbered circles that are randomly printed on a sheet of paper. In the CTT-2, numbered circles of 1 to 25 are shown twice (printed in pink and in yellow) randomly on a sheet of paper. Participants are asked to connect the numbers from 1 to 25 alternating between the two colors.
The changes over time in the results of Stroop Color Word Test (SCWT) (from baseline to the end of intervention) | Two weeks
  Stroop Color Word Test (SCWT), Chinese version; was administered to measure selective attention and cognitive flexibility. SCWT is composed of three parts, each lasting for 45 seconds.
The changes over time in the results of Tower of London test (from baseline to the end of intervention) | Two weeks
  A neuropsychological test for the assessment of executive functioning specifically to detect deficits in planning, which may occur due to a variety of medical and neuropsychiatric conditions.
The change over time in the score of the Digit Symbol Substitution Test (DSST) (from baseline to the end of intervention) | Two weeks
  DSST is a performance based test of cognitive performance tapping into processing speed, executive function, and attention, with 90 s test period and possible score range 0 133 (See detail in the DSST manual attached).
The changes over time in indices of heart rate variability (HRV) (from baseline to the end of intervention) | Two weeks
  HRV indices represent autonomic functioning. ECG electrodes were placed on bilateral arms just below the elbows, with a ground electrode placed just above the right wrist bone. Lead I electrocardiogram of each patient was taken for 5 min after sitting and having a rest for 20 min in a soundproof, dim-lighted room with thermostatic control. At baseline and the end of intervention, HRV will be collected during rest. The ECG signals were acquired, stored, pre-processed according to the recommended procedures and processed by an HRV analyser (LR8Z11, Yangyin Corp., Taipei, Taiwan). The time domain of HRV is obtained: Standard deviation of NN intervals (SDNN). Power spectrum of HRV is quantified into the standard frequency-domain measurements including low-frequency power (LF, 0.04-0.15 Hz), high-frequency power (HF, 0.15- 0.40 Hz).
The changes over time in EEG absolute power and coherence (from baseline to the end of intervention) | Two weeks
  In a recliner in a dimly lit, electrically shielded room, patients' EEGs were recorded at baseline and the end of intervention by using the Neuro Prax® TMS/tDCS full-band DC-EEG system with 32 EEG Ag/AgCl electrodes in the standard 10-20 International placement. EEG will be collected during resting eye-opened (5min) and eye-closed (5min) conditions. Signals will be amplified in the dynamic input range of ± 140 mV at a resolution of 0.5 μV by using EEG amplifiers and stored for offline analyses. Eye or muscle artifacts were automatically detected and removed using NeuroPrax's built-in software.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, M.D., Principal Investigator — Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwa
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No